CLINICAL TRIAL: NCT07047846
Title: Bowen Technique Versus Dynamic Soft Tissue Mobilization on Pain, Range of Motion and Functional Disability in Patients With Adhesive Capsulitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Collaborators: University of Lahore Hospital (ULH) (Network)
Responsible Party: Principal Investigator, Nadia Rehman, Physical Therapist, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-/494/08/24; The University of Lahore (Other: The University of Lahore)
Record Dates: First submitted 2025-06-04; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive Capsulitis; Bowen Therapy; Dynamic Soft Tissue Mobilization; range of motion; Shoulder Pain; physiotherapy
MeSH Terms: conditions — Bursitis; Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bowen technique with routine physical therapy (Experimental): This group will receive bowen technique 3 moves with routine physical therapy including ROM exercises, stretching exercises, strengthening exercises and scapular stabilization exercises . This group will receive 12 sessions ( 3 sessions per week)
  Interventions: Other: Bowen Technique and 3 moves
- Dynamic soft tissue mobilization with routine physical therapy (Active Comparator): This group will receive dynamic soft tissue mobilization with routine physical therapy including heat application , ROM exercises, stretching exercises, strengthening exercises and scapular stabilization exercises . This group will receive 12 sessions ( 3 sessions per week)
  Interventions: Other: Dynamic soft tissue mobilization

INTERVENTIONS:
Other: Dynamic soft tissue mobilization — Begin with gentle heat application or light massage to warm up the tissue for 5 minutes. Assess the range of motion and identify specific areas of tightness and pain. - Use hands or specialized tools to apply sustained pressure to the fascia and underlying muscles, concentrating on the scapular, pectoral, deltoidal, and rotator cuff muscles. Apply specific DSTM techniques to the identified muscles, gradually increasing the intensity as tolerated by the patient. Follow up with gentle stretching and strengthening exercises to maintain the gained ROM and improve muscle function.For subscapular are release Gentle circular movements over the subscapularis region to decrease the tension and increase the freedom of this muscle.For Supraspinatus and Infraspinatus Work Specific exercise over these muscles to help relieve pain and improve the shoulder joint.
  Arms: Dynamic soft tissue mobilization with routine physical therapy
Other: Bowen Technique and 3 moves — As the client sits, take a position across from the shoulder that needs attention. Hold the side you are working on by its forearm. Arrange the forearm so that it is horizontal at about chest level, keeping the elbow at a 90˚ angle and the shoulder apart from the trunk. Move 1: This is an anterior move that involves placing the fingers of the other hand over the midpoint of the triceps and posterior deltoid tendon, which is situated deeper. The ideal way to execute the exercise is to adduct the shoulder joint to its maximum ROM while placing the thumb of the same hand on the humeral head.Move 2: After the shoulder has fully adducted to the other side, strike the humeral head percussionally in the neck's direction. Move 3: Put the arm back in the beginning position and work the anterior deltoid at its midpoint with a supero-lateral move. Then take a pause for 2 minutes and repeat the moves. Complete 3 sets of all these moves in 35 minutes including 2 minutes pause after these 3 moves.
  Arms: Bowen technique with routine physical therapy

SUMMARY:
A randomized controlled trial included 72 patients diagnosed with adhesive capsulitis will conduct in University of Lahore Teaching Hospital. The study will complete within 9 months after the approval of synopsis. Patients who fulfilled the inclusion criteria will identified by individual physiotherapist and will enrolled for particular study. Informed written consent will be taken by the patients and will randomly allocated into two groups. The total numbers of sessions will 12 (3 sessions per week). The study will single blinded. The assessor will unaware of the treatment given to both groups.

Control group received routine physical therapy with dynamic soft tissue mobilization technique.

thermotherapy, trans-cutaneous electrical nerve stimulation, shoulder isometrics and stretching that includes 12 sessions and three times per week. Experimental group received routine physical therapy along with Bowen technique. This includes thermotherapy, trans-cutaneous electrical nerve stimulation, shoulder isometrics and stretching that includes 12 sessions and three times per week

DETAILED DESCRIPTION:
A randomized controlled trial will conduct at the UOL Teaching Hospital. Seventy-two diabetic patients aged 50-80 years with Grade 2 or 3 adhesive capsulitis will be divided into two groups at random: Bowen therapy will administered to Group A with routine physiotherapy, and Group B received DSTM with routine physiotherapy. Both interventions will delivered twice weekly for six weeks. Pain (VAS and SPADI Pain), ROM (flexion, abduction, external rotation), as well as functional impairment (SPADI Disability and Total Score) wil be assessed at baseline, week 3, and week 6.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed patients of 50-80 years of age
* Grade 2 & 3 (frozen and thawing) adhesive capsulitis
* patients willing to participate in the study
* Only diabetic patients

Exclusion Criteria:

* Major mental health probleme
* Patients who has a history of surgery on the shoulder, other shoulder diseases including a rotator cuff tear, sub acromial impingement syndrome, and a shoulder labral tear
* Patients taking oral or intra-articular steroids and cortisone injection prior 3 months
* Subjects with rotator cuff tears or other shoulder ligament injuries, H/O arthritis related to shoulder, malignancy, adhesive capsulitis secondary to fractures, dislocation, reflex sympathetic dystrophy, neurological disorder

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-07-16 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2026-01-03 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analogue Scale score | Change from preintervention to 6th weeks
  Visual analogue scale will be used to assess shoulder pain. Score ranges from 0-10. 0 shows least pain and 10 shows worst pain
Change in Universal Goniometer readings | Change from preintervention to 6th weeks
  Universal Goniometer will be used to assess shoulder range of motion.
change in Shoulder pain and disability Index (SPADI) | Change from preintervention to 6th weeks
  The 13 items of the SPADI measure two domains: an 8-item subscale measuring disability and a 5-item subscale measuring pain. The SPADI is available in two variants. The first version uses a visual analogue scale (VAS) to evaluate each item, while the second version uses a numerical rating scale (NRS).

CONTACTS AND LOCATIONS:
Locations (1):
- UOL Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hansen C, Taylor-Piliae RE. What is Bowenwork(R)? A systematic review. J Altern Complement Med. 2011 Nov;17(11):1001-6. doi: 10.1089/acm.2010.0023. PMID 22087611
- [Background] Aggarwal A, Saxena K, Palekar TJ, Rathi M. Instrument assisted soft tissue mobilization in adhesive capsulitis: A randomized clinical trial. J Bodyw Mov Ther. 2021 Apr;26:435-442. doi: 10.1016/j.jbmt.2020.12.039. Epub 2020 Dec 31. PMID 33992280
- [Background] Jusdado-Garcia M, Cuesta-Barriuso R. Soft Tissue Mobilization and Stretching for Shoulder in CrossFitters: A Randomized Pilot Study. Int J Environ Res Public Health. 2021 Jan 12;18(2):575. doi: 10.3390/ijerph18020575. PMID 33445505
- [Background] Carter B. A pilot study to evaluate the effectiveness of Bowen technique in the management of clients with frozen shoulder. Complement Ther Med. 2001 Dec;9(4):208-15. doi: 10.1054/ctim.2001.0481. PMID 12184347